CLINICAL TRIAL: NCT06542900
Title: Effectiveness and Safety of Deep Brain Stimulation(DBS) in Treatment-Resistant Depression(TRD)
Brief Title: Efficacy of Deep Brain Stimulation(DBS) for Treatment-Resistant Depression(TRD)
Acronym: DBS for TRD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBS for TRD
Record Dates: First submitted 2024-01-29; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-01

CONDITIONS: Treatment Resistant Depression
Keywords: TRD, DBS
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Treatment-Resistant Depression (TRD) (Experimental): Patients will undergo bilateral DBS lead implantation.
  Interventions: Device: Deep Brain Stimulation (DBS)

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) — The DBS lead is stereotactically introduced into the target in the brain (SCC, VC/VS, ALIC, ITP, NAc, LHb, MFB, or other unreported nuclei targets) and fixed to the skull; the lead is then connected to a neurostimulator implanted subcutaneously in the subclavicular region.

SUMMARY:
The primary purpose of this study is to investigate the effect of deep brain stimulation (DBS) implantation in patients with Treatment-resistant Depression (TRD) targeting the ventral capsule/ventral striatum (VC/VS), Brodmann area 25/subcallosal cingulate (SCC), Anterior Limb of Internal Capsule (ALIC), inferior thalamic peduncle (ITP), nucleus accumbens (NAc), lateral habenula (LHb), medial forebrain bundle (MFB), or other unreported nuclei targets.

DETAILED DESCRIPTION:
At least 40-60% of people with major depressive disorders (MDD) continue to have symptoms after treatment. The pharmacology treatment cannot produce sustained antidepressant effects in 50% of patients with depression. Therefore, more effective therapeutic methods are urgently needed. In a comprehensive survey of diverse neuromodulation therapies, targeting specific nuclei with deep brain stimulation (DBS) has the most potential for Treatment-resistant Depression (TRD) with apparent symptoms. The stimulation targets of DBS for patients with obsessive-compulsive disorder include the ventral capsule/ventral striatum (VC/VS), Brodmann area 25/subcallosal cingulate (SCC), Anterior Limb of Internal Capsule (ALIC), inferior thalamic peduncle (ITP), nucleus accumbens (NAc), lateral habenula (LHb), and medial forebrain bundle (MFB). However, the DBS case reports are limited and lack high-quality, evidence-based medical evidence. So, this cohort study focuses on the effectiveness of DBS-targeted VC/VS, SCC, ALIC, ITP, NAc, LHb, MFB, or other unreported nuclei targets on TRD.

Another goal of this program is to study the neuronal activity of the VC/VS, SCC, ALIC, ITP, NAc, LHb, MFB, or other unreported nuclei targets, respectively. At the same time, some subjects are presented with a task involving an unexpected reward. This separate study is an option and will not affect current study participation.

Some participants will also be invited to join a related study that involves positron emission tomography (PET) scanning to determine how the stimulation changes activity in the brain. Participation in the separate PET study is optional and will not affect current study participation.

ELIGIBILITY:
Inclusion Criteria:

1. male or female, 18-65 years old;
2. able to provide written informed consent voluntarily;
3. had a diagnosis of major depression disorder (MDD) (recurrent episodes) without psychotic features in compliance with the Diagnostic and Statistical Manual of Mental Disorders -Fourth Edition -Text Revised (DSM-IV-TR) and confirmed by the Mini-International Neuropsychiatric Interview Chinese version 5.0;
4. failure of response to at least two antidepressant medication trials based on the Massachusetts General Hospital antidepressant treatment response questionnaire (MGH-ATRQ);
5. ongoing antidepressant(s) at a fixed dose for at least four weeks before baseline assessment;
6. had a score of ≥201 on the Hamilton Depression Scale- item 17 (HAMD-17) at baseline.

Exclusion Criteria:

1. presence of other psychotic disorders;
2. have a treatment history that includes electroconvulsive therapy (ECT), modified electroconvulsive therapy (MECT), transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), DBS, and transcranial magnetic stimulation (TMS);
3. presents a suicide risk (defined as a HAMD-17 score of ≥3 on suicide-related items);
4. experience difficulty in effectively communicating with investigators;
5. with a history of traumatic brain injury (TBI);
6. with intracranial or cardiovascular stents;
7. substance abuse within the past six months;
8. unstable neurological or coagulation disorders;
9. women who are pregnant, lactating, or of childbearing potential who refuse the use of reliable contraception during the study;
10. have been involved in other clinical studies within three months before enrollment in this study;
11. any conditions considered by the study group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The change from baseline to 12 months in the Montgomery-Asberg Depression Rating Scale (MADRS) total score. | Baseline to 12 months post-surgery
  MADRS is an established instrument to rate symptoms of depression. The range of the total score is thus 0 to 60; higher total scores indicate more severe depressive symptoms.
  Usual cutoff points are: 0 to 6: normal/symptom absent; 7 to 19: mild depression; 20 to 34: moderate depression; >34: severe depression.

SECONDARY OUTCOMES:
Remission, and response rate at week 2, month 3, month 6, and month 12, revealed by Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline to week 2, month 3, month 6, and month 12
  the Montgomery-Åsberg Depression Rating Scale (MADRS) score (range, 0 to 60, with higher scores indicating more severe depression.
  Remission and response were defined as a MADRS score ≤10 and a >50% reduction from the baseline MADRS score, respectively.
the change from baseline to 2 weeks, 3 months, 6 months, and 12 months in the Hamilton Anxiety Rating Scale (HAMA) total score. | Baseline to week 2, month 3, month 6, and month 12
  HAMA is a 14-item test measuring the severity of anxiety symptoms. The total anxiety score ranges from zero to 56, with higher scores indicating more anxiety. The seven psychic anxiety items elicit a psychic anxiety score that ranges from 0 to 28. The remaining seven items yield a somatic anxiety score ranging from 0 to 28.
the changes of Hamilton Depression Rating Scale, 17 item (HAMD-17) scores and its subscales from baseline to 2 weeks, 3 months, 6 months, and 12 months. | Baseline to week 2, month 3, month 6, and month 12
  HAMD-17 ranges from 0 to 52, with higher scores indicating more depression; a score of 20 or more indicates moderate to severe depression.
the change of Pittsburgh Sleep Quality Index (PSQI) from baseline to Week 2, Month 3, Month 6, and Month 12. | Baseline to week 2, month 3, month 6, and month 12
  PSQI is a 19 items measurement of several aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
the change from baseline to 2 weeks, 3 months, 6 months, and 12 months in Clinical Global Impression-Severity scale (CGI-S) | Baseline to week 2, month 3, month 6, and month 12
  The Clinical Global Impression-Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment. Score 1 presents normal, not at all ill, and score 7 presents among the most extremely ill patients.
the change of Clinical Global Impression-Improvement scale (CGI-I) at Week 2, Month 1, Month 3, Month 6, and Month 12. | Baseline to week 2, month 3, month 6, and month 12
  The Clinical Global Impression-Improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Score 1 presents the patient as much improved, and score 7 presents much worse.
the change from baseline to Week 2, Month 3, Month 6, and Month 12 in EuroQol-5 Dimension-level Scale (EQ-5D-5L). | Baseline to week 2, month 3, month 6, and month 12
  EQ-5D-5L is an instrument that evaluates the generic quality of life. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The score ranges from 5 (having no problems) to 25 (being unable to do/having extreme problems).
the change from baseline to Week 2, Month 1, Month 3, Month 6, and Month 12 in Young Mania Rating Scale (YMRS). | Baseline to week 2, month 3, month 6, and month 12
  This scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. Scores range from 0 to 60, with higher scores indicating more severe mania. A score of 0 to 5 means no obvious manic symptoms; a score of 6 to 10 means definite manic symptoms; a score of 22 or above means severe manic symptoms. It will be used as a systematic screen for DBS-induced mania or hypomania. Although scores above 8 have been considered evidence of manic symptomatology in bipolar patients, the unmasked physician will use this scale and screening questions to assess whether any hypomanic symptoms require clinical intervention including DBS adjustment.
Safety as indicated by the number of Adverse Events at Week 2, Month 3, Month 6, and Month 12. | Baseline to week 2, month 3, month 6, and month 12
  Possible Adverse Events include:
  Major and minor adverse events will be evaluated by Adverse Events Questionnaire (AEQ) and accompanying Case Report Form (AEQ CRF) in multiple domains, including psychiatric, neurological, and cognitive effects. The AEQ includes cognitive and behavioral screening items used in the Xuanwu DBS clinic for movement disorder patients. Additionally, we have added items for the adverse events observed in pilot DBS for TRD.
the change from baseline to Month 12 in the Controlled Oral Word Association Test (COWAT). | 1 year after neurostimulator implantation.
  During the Controlled Oral Word Association Test (COWAT), individuals are tasked with verbally generating words starting with different letters of the alphabet. They have 60 seconds for each letter to retrieve and articulate as many words as possible. The test involves presenting three letters, each progressively more challenging in associative difficulty. Scores are derived by summing the total words produced across the three letter trials. The lowest achievable score is zero, indicating an inability to generate any words. There is no upper limit to the score as participants can produce numerous words for each letter. Higher scores reflect superior word retrieval and cognitive function.
the change from baseline to Month 12 in the Trail-Making Test A&B | 1 year after neurostimulator implantation.
  The Trail-Making Test A and B assess cognitive shifting, visual search speed, scanning, processing speed, mental flexibility, and executive functioning. It evaluates the participant's capacity for sequencing (Parts A and B), cognitive set shifting (Part B), and processing speed (Parts A and B). Scores for Part A and Part B are calculated independently, indicating the number of seconds required for the participant to finish each section. Higher scores denote longer durations for completing the test.
the change from baseline to Month 12 in Rey-Osterrieth Complex Figure Test (ROCF). | 1 year after neurostimulator implantation.
  The Rey-Osterrieth complex figure test (ROCF) is a neuropsychological assessment in which patients are asked to reproduce a complicated line drawing, first by copying it freehand (recognition), and then drawing from memory (recall). Scoring of drawings is based on the widely used 36-point scoring system (0 being the worst score and 36 the best).

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Wang, MD & PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided